CLINICAL TRIAL: NCT05142072
Title: Formulation, Characterization and In-vivo Evaluation of Controlled Release Intranasal Films of Vitamin D3 as an Optimistic Dosage Form for Rapid and Effective Healing of Cauterized Turbinectomy
Brief Title: Design and Application of Vitamin D Films for Burn Healing After Cauterizing Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Deraya University (Other)
Responsible Party: Principal Investigator, Soad Ali, lecturer of pharmaceutics and clinical pharmacy Deraya university, Deraya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DNFs; Ahmed Ali (Other: minia university faculty of medicine)
Record Dates: First submitted 2021-10-25; First posted 2021-12-02 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Nasal Obstruction
MeSH Terms: conditions — Nasal Obstruction | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vitamin D film (Experimental): Prepared intranasal films containing vitamin D3 by the investigators and administered to the right nostril with the aid of an ENT surgeon
  Interventions: Drug: Vitamin D3
- control group (Other): No devices will be added
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — intranasal film
  Other Names: Calciferol

SUMMARY:
One of this method's drawbacks is the healing of cauterized cartilage after processing. It was reported that the healing is so slow as no dosage form can reach this place in addition to the scares produced from healing is very irritable to the patient.

From this point, the investigators start searching for a solution to this problem and reach the repositioning of Vitamin D3 (calciferol) as an active ingredient for the rapidity and efficacy of burn healing.

The dosage form of choice that was reported before for intranasal application by the same team of investigators and gave good results. the intranasal films were proved for its convince, simplicity, efficacy, and compliance to patients.

ELIGIBILITY:
Inclusion Criteria:

* patients complain of nasal obstruction
* do not respond to medications
* treatment need surgery
* patients accept following up in a timely manner for 3 weeks

Exclusion Criteria:

* no nasal polyps,
* have problems with the surgical procedures
* have allergy with any of the treatment components (vitamin D3 or chitosan)
* don't follow instructions or miss the following up

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-12-18 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
Healing of cauterized tissues after surgery procedures | three week
  The outcome will be measured by endoscopic scanning pre and after application of the drug in the dosage form (representing the percent of healing) by the ENT surgeon.

SECONDARY OUTCOMES:
patients compliance from the new dosage form | three weeks
  The patient compliance will be measured by rating the pain and the development of symptoms before surgery using a questionnaire
Assessment of grades of healing by ENT surgeon | three weeks
  Evaluation of (1) bleeding (amount and frequencies), (2) crustation ( amount and nature), and (3) inflammation (size and the redness of the place of surgery)

CONTACTS AND LOCATIONS:
Locations (1):
- Minya university, faculty of medicin, Minya, Minya Governorate, Egypt